CLINICAL TRIAL: NCT05829798
Title: An Efficacy and Safety 6-months Study of SYNOLIS VA 80/160 and SYNOLIS VA 40/80 in the Treatment of Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aptissen SA (Industry)
Collaborators: Noblewell (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMCF2-4ML single injection
Record Dates: First submitted 2023-03-21; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee Osteoarthritis; Hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYNOLIS VA 80/160 (Experimental): SYNOLIS VA 80/160 (hyaluronic acid 80 mg, sorbitol 160 mg) Intra-articular injection
  Interventions: Device: SYNOLIS VA 80/160
- SYNOLIS VA 40/80 (Experimental): SYNOLIS VA 40/80 (hyaluronic acid 40 mg, sorbitol 80 mg) Intra-articular injection
  Interventions: Device: SYNOLIS VA 40/80

INTERVENTIONS:
Device: SYNOLIS VA 80/160 — Single 4mL intra-articular injection of SYNOLIS VA 80/160
  Arms: SYNOLIS VA 80/160
Device: SYNOLIS VA 40/80 — Single 2mL intra-articular injection of SYNOLIS VA 40/80
  Arms: SYNOLIS VA 40/80

SUMMARY:
Multicentre, independent assessment study on SYNOLIS VA 80/160 and SYNOLIS VA 40/80 over a period of 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patient between 35 and 75 years old
* Patients with knee osteoarthritis. The diagnosis is based on the following American College of Rheumatology (ACR) classification:

  * Knee pain
  * Positive radiography (presence of osteophytes)
  * Morning stiffness < 30 min and/or crepitus while walking
* Symptoms related to knee osteoarthritis for at least 6 months
* Treatment failure (i.e. ineffective response) with analgesics and/or NSAIDs or intolerance to NSAIDs or low-grade opioids
* Kellgren-Lawrence radiographic stage: I - III (pre-inclusion radiography)
* WOMAC pain index score ≥ 40 mm (VAS 0-100 mm) on the knee to be treated
* Contralateral knee pain < 10 mm (VAS) compared to treated knee
* Patient signed inform consent form-

Exclusion Criteria:

* Inability to understand the study or language used to be informed/sign the consent
* Participation in another clinical trial within 4 weeks prior to the start of the trial, and commitment to non-participation within 4 weeks following the end of the trial
* Intraarticular injection of hyaluronic acid in target knee within the 6 months prior to inclusion
* Patient who has received an intra-articular (IA) or intra-muscular (IM) steroid injection within the 3 months prior to inclusion or has taken oral corticosteroids within the month prior to inclusion
* Joint, bone, ligament, or any local or loco-regional surgery of the leg involved, arthroscopic operation on the target knee within the 3 months prior to inclusion
* Any recent trauma to the leg involved, including a sprain, dislocation within the 3 months prior to inclusion
* Rheumatoid arthritis, joint condition or any other inflammation and arthritis
* Lupus
* Dermatological disorder or any epidermal conditions that prevent an intraarticular injection
* Visible joint effusion of the target knee during physical examination evidenced by a protuberance or positive ballottement of the patella
* Evidence of a subchondral fracture, meniscal lesion, presence of bone or cartilage fragments, horizontal meniscal lesion tear (FLAP) in the target knee
* Osteonecrosis (1 or both knees)
* Daily dosage > 101 mg of acetylsalicylic acid as part of cardiovascular preventive treatment (antithrombotic). If dose < 101 mg, must be maintained during the study
* Known intolerance/hypersensitivity/allergy to any of the components in either product, SYNOLIS VA
* Fibromyalgia
* Patient of childbearing potential, pregnant or breast-feeding known at inclusion or in the planning phase during the study unless willing to use contraceptives through the whole duration of the study
* Excessive and repeated consumption of alcohol or illicit substances
* Any medical condition that may interfere with the proper conduct of the study (including any surgery or hospitalisation)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Difference in Western Ontario and McMaster Universities Arthritis index (WOMAC) score total between D168 and inclusion visit | 168 days
  The Western Ontario and McMaster Universities Arthritis index (WOMAC) is a 24-item, condition-specific questionnaire available in a 5-point Likert and 100 mm visual analog scale (VAS) as well as an 11-box numerical rating scale, composed of three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). VAS was used in this study, with a score of 0 for no pain and 100 mm for the worst pain one can image)

SECONDARY OUTCOMES:
Change in pain measurements, assessed using the Western Ontario and McMaster Universities Arthritis index (WOMAC) pain severity index, as compared to D0 | up to 168 days
  The Western Ontario and McMaster Universities Arthritis index (WOMAC) is a 24-item, condition-specific questionnaire available in a 5-point Likert and 100 mm visual analog scale (VAS) as well as an 11-box numerical rating scale, composed of three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). VAS was used in this study, with a score of 0 for no pain and 100 mm for the worst pain one can image)
Change in the Western Ontario and McMaster Universities Arthritis index (WOMAC) functional severity index, as compared to D0 | up to 168 days
  The Western Ontario and McMaster Universities Arthritis index (WOMAC) is a 24-item, condition-specific questionnaire available in a 5-point Likert and 100 mm visual analog scale (VAS) as well as an 11-box numerical rating scale, composed of three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). VAS was used in this study, with a score of 0 for no pain and 100 mm for the worst pain one can image)
Change in the Western Ontario and McMaster Universities Arthritis index (WOMAC) stiffness severity index, as compared to D0 | up to 168 days
  The Western Ontario and McMaster Universities Arthritis index (WOMAC) is a 24-item, condition-specific questionnaire available in a 5-point Likert and 100 mm visual analog scale (VAS) as well as an 11-box numerical rating scale, composed of three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). VAS was used in this study, with a score of 0 for no pain and 100 mm for the worst pain one can image)
Percentage of subjects using analgesics | up to 168 days
  New NSAID / analgesics drugs usage
Measurement of relief satisfaction by the patient | 168 days
  7-point Likert scale (1 point very unsatisfied to 7 points for very satisfied)
Measurement of therapeutic efficacy by the investigator (assessor) | 168 days
  7-point Likert scale (1 point very unsatisfied to 7 points for very satisfied)

OTHER OUTCOMES:
Safety and tolerability of SYNOLIS VA 80/160 and SYNOLIS VA 40/80 assessed with adverse events monitoring throughout the study duration | 168 days

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - SPORTO Spółka z o.o., Lodz
  - Klinika Chirurgii Kolana Dr Słynarskiego, Warsaw
  - NZOZ Carolina Medical Center - Sport Medica S.A, Warsaw